CLINICAL TRIAL: NCT05783648
Title: Do Anesthesiologists Follow Guidelines on Perioperative Use of Tranexamic Acid?
Acronym: Periop_TXA
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SRB2023055
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-03

CONDITIONS: Tranexamic Acid; Blood Loss, Surgical; Blood Transfusion
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before TXA recommendations: All patients operated between october 1st, 2021 and december 31st 2021, that means before the publication of the POISE-3 trial and the recommendations on the use of tranexamic acid.
  Interventions: Drug: Use of tranexamic acid
- After TXA recommendations: All patients operated between october 1st, 2022 and december 31st 2022, that means after the publication of the POISE-3 trial and the recommendations on the use of tranexamic acid.
  Interventions: Drug: Use of tranexamic acid

INTERVENTIONS:
Drug: Use of tranexamic acid — Percentage of correct use according to POISE-3 criteria of tranexamic acid

SUMMARY:
Tranexamic acid has been used to reduce bleeding and transfusion for years. Randomized studies showed its efficacity in orthopedic surgery, trauma and post-partum hemorrhage. Few data were available for other types of surgery and the safety profile of tranexamic use was nor clearly established. In april 2022, the results from the POISE-3 (Perioperative Ischemic Evaluation - 3) trial was published in the New England Journal of Medicine. This stdy clearly demonstrated in 9535 patients undergoing non-cardiac surgery, that the use of tranexamic acid significantly reduced not only perioperative bleeding, but also transfusions. The safety profile of tranexamic acid was very good in this trial. This publication was rapidly followed by editorials in major anesthesia journals, calling for "safe surgery" with a systematic use of tranexamic acid in the population studied in the POISE-3 trial. A literature review was done with a formal presentation at Erasme University Hospital, again with the call for a systematic use in appropriate patients.

In this study, the adherence to these recommendations will be tested. All patients operated between october 1st 2022 and december 31 st 2022 will be included. For every patient, it will be determined if this patient should have received tranexamic acid according to the results of the POISE-3 trial and wether this patient really did get tranexamic acid. Primary endpoint will be the percentage (%) of patients correctly treated according to the POISE-3 recommendations. A second primary endpoint will be the comparison with patients operated between October 1st 2021 and december 31st 2021; that means before the publication of the recommendations. The difference between both populations will be tested with a Chi-square test. Secondary outcomes wil be bleeding and transfusion in the correctly treated population compared with an eventually not correctly treated population.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery either between oct 1st 2021 and dec 31st 201 or oct 1st 2022 and dec 31st 2022
* noncardiac surgery
* expected to require at least one overnight hospital admission after surgery
* at risk of perioperative bleeding

Exclusion Criteria:

* cardiac surgery
* intracranial neurosurgery
* creatinine clearance < 30 mL/min (Cockcroft-Gault equation)
* chronic dialysis
* history of seizure disorder
* recent (< 3 months) stroke, myocardial infarction, acute arterial thrombosis, venous thromboembolism
* fibrinolytic condition following consumption coagulopathy
* subarachnoid hemorrhage within 30 days before surgery
* women of childbearing potential who are not taking effective contraception, pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing inpatient surgery either between oct 1st 2021 and dec 31st 2021 or oct 1st 2022 and dec 31st 2022
Sampling Method: Non-Probability Sample
Enrollment: 1726 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Percentage of correct use of TXA | 12 hours
  Percentage of patients who received tranexamic acid correctly according to the POISE-3 criteria
Comparison of percentage use of TXA before and after the release of TXA recommendations | 12 hours
  The use of tranexamic acid (in percentage) will be compared between the two cohorts, before and after the publication of the recommendations on the use of tranexamic acid

SECONDARY OUTCOMES:
Blood loss | 24 hours
  Comparison of blood loss between correctly treated patients and not correctly treated patients according to the POISE-3 criteria
Transfusion | 24 hours
  Comparison of blood transfusion between correctly treated patients and not correctly treated patients according to the POISE-3 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Universitaire de Bruxelles - Hôpital erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No